CLINICAL TRIAL: NCT03687333
Title: A Single Arm, Prospective, Open-label, Multi-center Study to Evaluate Efficacy and Safety in Chinese Patients With Infantile-Onset Pompe Disease With One Year Alglucosidase Alfa Treatment
Brief Title: Evaluate Efficacy and Safety in Chinese Patients With Infantile-Onset Pompe Disease With One Year Alglucosidase Alfa Treatment
Acronym: APOLLO-IOPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALGMYL08718; U1111-1203-8484 (Other: UTN)
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alglucosidase Alfa therapy (Experimental): Alglucosidase Alfa dose is calculated per kg body weight and administered once every 2 weeks for up to 52 weeks.
  Interventions: Drug: ALGLUCOSIDASE ALFA (MYOZYME)

INTERVENTIONS:
Drug: ALGLUCOSIDASE ALFA (MYOZYME) — Pharmaceutical form: cake or powder for injection
  Route of administration: intravenous infusion

SUMMARY:
Primary Objective:

To evaluate effect of 52-week treatment with Alglucosidase Alfa in the extension of survival and improvement of cardiomyopathy measured by Left Ventricular Mass Index in Chinese patients with infantile-onset Pompe Disease.

Secondary Objectives:

* To observe the improvement of physical growth, motor and cognitive development of 52-week treatment with Alglucosidase Alfa in infantile-onset Pompe Disease from the baseline.
* To observe the efficacy on survival free of invasive ventilation, use of any ventilation support of 52- week treatment with Alglucosidase Alfa in Chinese patients with infantile-onset Pompe Disease.
* To evaluate the safety and tolerability of Alglucosidase Alfa in Chinese patients with infantile-onset Pompe Disease.

DETAILED DESCRIPTION:
Total of 56 weeks in the study period, including an up to 28-day screening period and 52-week treatment period, followed by 30-day post-treatment observation period.

After the end of 52-week treatment, patients' guardians could choose to participate in a patient assistance program (PAP) sponsored by Sanofi and launched before first patient out (FPO) or reimbursement from social insurance for continued treatment.

ELIGIBILITY:
Inclusion criteria:

* Subject's parents or legal guardians must provide written informed consent prior to any study-related procedures.
* Documented onset of Pompe disease symptoms up to 12 months of age (corrected for gestation if born before 40 weeks); diagnosis of Pompe disease confirmed by acid alpha-glucosidase enzyme deficiency from any tissue source and acid alpha-glucosidase gene mutations.
* Age 0-12 months at enrollment, defined as at the time of providing written informed consent.
* Cardiomyopathy (abnormal left ventricular mass indices [LVMIs], measured by echocardiography, abnormal value is defined as ≥65 g/m2 for patients up to 12 months old) confirmed by cardiologist at study site.

Exclusion criteria:

* Patient who has previously been treated with acid alpha-glucosidase.
* Patient who is participating in another clinical study using any investigational therapy.
* Conditions/situations such as:
* Clinical signs of cardiac failure with ejection fraction < 40%.
* Respiratory insufficiency (oxygen saturation < 90% or carbon dioxide partial pressure > 55 mm Hg [venous] or > 40 mm hydrargyrum [arterial] in room air or any ventilator use).
* Patients who are dependent on invasive or non-invasive ventilator support.
* Patients with major congenital anomaly or clinically significant intercurrent organic disease unrelated to Pompe disease.
* Patients not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or patients potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Survival | at week 52
  The proportion of patients alive at the end of study
Left Ventricular Mass Index (LVMI) | at week 52
  Change from baseline in LVMI

SECONDARY OUTCOMES:
Invasive ventilation-free survival | at week 52
  Survival free of invasive ventilator use at 52-week treatment
Any ventilation-free survival | at week 52
  Survival free of any ventilator use at 52-week treatment
Growth in body weight and length | at week 52
  Physical growth: Change from baseline at Week 52 with regards to length and weight
Motor development milestones | at week 52
  Number of motor development milestones achieved at Week 52 and change from baseline
GESELL Development Scale | at week 52
  Change from baseline at Week 52 on GESELL Developmental Scale
Cardiac failure | at week 52
  Proportion of patients with signs and/or symptoms of cardiac failure at Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site number, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Zhu D, Zhu J, Qiu W, Wang B, Liu L, Yu X, Ou Z, Shan G, Wang J, Li B, Chen X, Liu C, Li Z, Fu L. A Multi-Centre Prospective Study of the Efficacy and Safety of Alglucosidase Alfa in Chinese Patients With Infantile-Onset Pompe Disease. Front Pharmacol. 2022 Jun 27;13:903488. doi: 10.3389/fphar.2022.903488. eCollection 2022. PMID 35833019